CLINICAL TRIAL: NCT02346825
Title: Multisite RCT of 3 Neurorehabilitation Therapies for Infants With Asymmetrical Cerebral Palsy
Brief Title: The Baby CHAMP Study (Children With Hemiparesis Arm and Movement Project)
Acronym: The Baby CHAMP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Ohio State University (Other); University of Virginia (Other)
Responsible Party: Principal Investigator, Stephanie DeLuca, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01HD074574-01A1 (NIH)
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Hemiparesis; Cerebral Palsy
Keywords: P-CIMT; Pediatric Constraint Induced Movement Therapy; Hemiparesis; Cerebral Palsy; Infants; Toddlers; Children
MeSH Terms: conditions — Paresis; Cerebral Palsy | interventions — POLR1G protein, human; Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intensive Plus Cast (Experimental): Children in this group will have 3 hours of daily therapy each weekday for 4 weeks while wearing a full-arm cast on their stronger arm and hand. Parents will be required to do 45 minutes of daily therapy for which they will be trained.
  Interventions: Behavioral: Neurorehabilitation therapy with cast
- Intensive Plus Splint (Experimental): Children in this group will have 3 hours of daily therapy each weekday for 4 weeks while wearing a part-time splint on their stronger arm and hand. Parents will be required to do 45 minutes of daily therapy for which they will be trained.
  Interventions: Behavioral: Neurorehabilitation therapy with splint
- Intensive no Constraint (Experimental): Children in this group will have 3 hours of daily therapy each weekday for 4 weeks but will not wear a constraint. Parents will be required to do 45 minutes of daily therapy for which they will be trained.
  Interventions: Behavioral: Neurorehabilitation bimanual

INTERVENTIONS:
Behavioral: Neurorehabilitation therapy with cast — Children in this group will have 3 hours of daily therapy each weekday for 4 weeks while wearing a full-arm cast on their stronger arm and hand. Parents will be required to do 45 minutes of daily therapy for which they will be trained.
  Other Names: Pediatric Constraint-Induced Movement Therapy; P-CIMT
  Arms: Intensive Plus Cast
Behavioral: Neurorehabilitation therapy with splint — Children in this group will have 3 hours of daily therapy each weekday for 4 weeks while wearing part-time splint on their stronger arm and hand. Parents will be required to do 45 minutes of daily therapy for which they will be trained.
  Other Names: Pediatric Constraint-Induced Movement Therapy; P-CIMT
  Arms: Intensive Plus Splint
Behavioral: Neurorehabilitation bimanual — Children in this group will have 3 hours of daily therapy each weekday for 4 weeks will not wear a constraint. Parents will be required to do 45 minutes of daily therapy for which they will be trained.
  Other Names: Bimanual; HABIT
  Arms: Intensive no Constraint

SUMMARY:
The Baby CHAMP Study is a multisite clinical trial funded by the National Institutes of Health that is examining the the use of constraint-induced movement therapy (CIMT) for infants and toddlers as a effective treatment, since there have been no randomized control trials (RCT) for the age range as well as monitor the stress levels as related by self-report of parents or biological indicators. Infants and toddlers who meet study eligibility requirements at one of the three clinical sites (Charlottesville, VA, Columbus, OH, and Roanoke, VA) will be invited to enroll, and their parents will be provided all necessary paperwork along with informational documentation.

DETAILED DESCRIPTION:
In 2013, a systematic review of interventions for children with cerebral palsy (Novak et al, 2013) concluded that constraint-induced movement therapy (CIMT) produces the largest magnitude effects of any non-surgical treatment. Similarly, the first major handbook summarizing the results from more than 50 studies on CIMT conducted worldwide (Ramey, Coker-Bolt, & DeLuca, 2013) provides additional clinical and scientific support for the conclusion that CIMT can produce significant benefits. There are a number of important unresolved issues. One concerns the need for empirical evidence that CIMT is efficacious for infants and toddlers, since there has been no randomized controlled trial (RCT) focused on this age range. Another issue under debate is whether there are different effects related to the type of constraint used during the therapy. The constraint is placed on the child's "stronger" or non-hemiparetic upper extremity while the therapy focuses on improving the child's skills in using the impaired or hemiparetic upper extremity. Two widely used forms of constraint are: 1) a full-arm cast that the child wears continuously throughout a multi-week period when the child receives daily therapy and 2) a part-arm splint that the child wears only during the time of day when he or she receives therapy. Finally, another important topic that has not been studied is whether CIMT is a stressful form of therapy, because it is high-intensity (i.e., much higher dosage than the usual and customary sessions in other forms of occupational and physical therapy), involves constraining the child's non-involved or less involved upper extremity, and takes place in the child's home and often asks parents to help with practice sessions during non-therapy hours. If CIMT does produce elevated stress for the child, the parents, or both, is this stress short-term (i.e., just at the start of therapy) or does this continues over the entire period of therapy? Further, does the type of constraint used produce different levels of stress, either at first or throughout the course of therapy?

The proposed study is a randomized controlled trial (RCT) of CIMT for 72 children with hemiparetic spastic cerebral palsy (CP) between the ages of 6 and 24 months. The study will take place in two sites (Roanoke, VA and Columbus, OH), each site enrolling 36 children over a 3 year period. The study will address two specific aims:

Aim 1: to test the efficacy of 3 different constraint conditions used as part of administering a standardized form of therapy known as ACQUIRE (DeLuca, Echols, & Ramey, 2007). The 3 constraint conditions are: i) continuous constraint, ii) part-time constraint, and iii) no constraint. In all 3 groups, children will receive 3 hours of therapy per day for 5 days per week for 4 consecutive days. Therapy is delivered by licensed occupation or physical therapists who have been trained to deliver ACQUIRE therapy to high fidelity. In addition, parents are trained to provide one hour of practice in their homes, using techniques compatible with those used by the ACQUIRE therapist. Efficacy will be measured primarily by changes in the children's assessed skill levels in using their upper extremities, both the hemiparetic (affected) and the non-hemiparetic (less involved) upper extremities, used alone and together (i.e., in completing bimanual tasks). In addition, changes in brain functioning related to receiving the 3 different constraint conditions will be measured using functional Near-Infrared Spectroscopy (fNIRS), a non-invasive and safe procedure that permits children to be active while recording takes place.

Aim 2: to monitor stress levels and safety risks related to use of constraint in the 3 conditions identified above (Aim 1). The study addresses stress levels in both the children and their parents, because CIMT is a high-intensity and unusual (i.e., constraining the child's "stronger arm") form of therapy taking place in the children's homes. Prior published clinical case reports indicate infants and toddlers adjust well to this form of therapy, and parents have favorable responses, no study previously has directly measured stress effects, related to self-report of parents or biological indicators, such as revealed by collecting saliva and hair samples to analyze for cortisol levels and changes over time.

The study results are expected to be important to inform the field of infant rehabilitation and provide much-needed evidence about whether infants and toddlers show significant (clinically meaningful) benefits from one or more of the 3 forms of therapy being tested. The findings will include evidence about both behavioral and brain changes. Further, the evidence will answer questions about whether the immediate therapy benefits, if detected, continue to be measurable at 6 and 12 months after therapy has ended. In addition, the study will yield first-ever evidence about whether CIMT is stressful for children and their parents. It may be there are some children or parents who are at higher risk for showing stress effects. If so, the data generated by this study will be important for future clinical practice and research to reduce these levels. If elevated stress does not occur, or if markedly lowering of stress is detected, then these findings will help to resolve the uncertainty that currently prevents some families or clinicians from considering this form of therapy, despite the fact that other scientific studies have shown it produces large and lasting benefits for children age 2 and older.

ELIGIBILITY:
Inclusion Criteria:

1. child is 6 - 24 months old
2. diagnosis of unilateral/asymmetrical Cerebral Palsy
3. has functional upper extremity impairment levels of II, III, or IV (Manual Abilities Classification System, Eliasson et al 2006)
4. parent(s) willing to be partners in study and participate in follow-up assessments for 12 mos.

Exclusion Criteria:

1. medical or sensory condition that prevents full therapy participation (e.g., frequent uncontrolled seizures, blindness)
2. received CIMT or had botulinum toxin therapy in past 6 mos.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in the Mini - Assisting Hand Assessment | immediatly prior to treatment, immediately after treatment, 6 months after treatment, 12 months after treatment
  functional assessment
Change in the Bayley Infant Scales of Development | immediatly prior to treatment, immediately after treatment, 6 months after treatment, 12 months after treatment
  functional assessment

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The Ohio State University, Columbus, Ohio
  - University of Virginia, Charlottesville, Virginia
  - Fralin Biomedical Research Institute at Virginia Tech, Roanoke, Virginia